CLINICAL TRIAL: NCT07161154
Title: Sentio Systematic Evaluation - SENSE
Brief Title: Sentio Systematic Evaluation
Acronym: SENSE
Status: Not yet recruiting | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BC125
Record Dates: First submitted 2025-07-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Bilateral or Unilateral; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Single Sided Deafness; Hearing Loss; Hearing-Impairment; Hearing Aid
Keywords: Active transcutaneous bone conduction hearing system
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sentio: Patients recieving the Sentio system
  Interventions: Device: Transcutaneous bone conduction hearing system

INTERVENTIONS:
Device: Transcutaneous bone conduction hearing system — The Sentio system is an active transcutaneous bone conduction hearing system (single armed study)

SUMMARY:
The study is designed as an international, multi-center, single-armed, non-interventional/observational study including subjects who has received or are planned to receive the Sentio system as part of normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject who is scheduled for or have undergone Sentio implantation in clinical practice.
* Subject who has consented to participation or are covered by consent waiver.

Exclusion Criteria:

* Subjects enrolled in other clinical investigations leading to their Sentio implantation and subsequent follow-up deviating substantially from clinical practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving the Sentio system in clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Rate of succesful use of the device | Completion of the surgical procedure is reported at the surgery. Device specific questionnaire is typically completed within the first year of follow-up, though timing may vary depending on local practice for follow-up.
  Successful use is defined as a composite outcome consisting of completion of the surgical procedure and patient reported satisfaction after fitting and use of the device (assessed through a device specific questionnaire).

SECONDARY OUTCOMES:
Frequency of surgical events and complications | During surgery
Assess surgical approaches and techniques | During surgery
Frequency of post-operative complications | From surgery till end of follow-up (expected up to 10 years)
Timing of fitting | During fitting appointment (typically 2-15 weeks after surgery, depending on patient needs and local variations on practice)
  Days between surgery and fitting of sound processor.
To assess improvement in hearing | At fitting and throughout follow-up period (expected up to 10 years)
  Free-field thresholds

IPD SHARING:
Plan to Share IPD: No
To protect integrity of patients.